CLINICAL TRIAL: NCT01328405
Title: The Air-Q Intubating Laryngeal Airway Versus the LMA-Proseal: A Prospective, Randomized Trial of Airway Seal Pressure
Brief Title: Air-Q Intubating Laryngeal Airway Versus the Laryngeal Mask Airway (LMA)-Proseal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2009-0012
Record Dates: First submitted 2011-03-29; First posted 2011-04-04 (Estimated); Results first posted 2012-08-10 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2012-07

CONDITIONS: Difficult Airway; Anesthesia; Functional
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air-Q LMA (Experimental): Air-QⓇ intubating laryngeal mask (Mercury Medical, Clearwater, Fl.)
  Interventions: Device: Laryngeal Mask Airway (LMA)
- Proseal LMA (Experimental): LMA-Proseal TM (LMA North America, San Diego, Ca.)
  Interventions: Device: Laryngeal Mask Airway (LMA)

INTERVENTIONS:
Device: Laryngeal Mask Airway (LMA) — Comparison of airway seal pressure, airway morbidity bronchoscopic view obtained between two different laryngeal mask airways.
  Other Names: Air-QⓇ intubating laryngeal mask(Mercury Medical,Clearwater, Fl.); LMA-Proseal TM(LMA North America,San Diego, Ca.)

SUMMARY:
Introduction:

The air-QⓇ Intubating Laryngeal Airway (ILA) is a newer supraglottic airway. It is approved for use as a primary airway and as an aid for intubation in situations of anticipated or unanticipated difficult airways. A unique feature of this device as compared to other airways on the market is the size of the inner diameter (ID) and length of its airway tube. Direct placement of tracheal tubes > 7.5 mm ID through the airway tube is possible.

The ProSealTM LMA is considered the gold standard for supraglottic devices with respect to airway seal pressure. On average, it is reported to be approximately 28 cmH2O. This is significantly higher than that of the first generation LMA, the LMA-ClassicTM, which has a maximum seal pressure of 20 cmH2O, but averages 16-18 cmH2O in actual practice.

In this study the investigators aim to test whether the air-QⓇ creates an airway seal pressure that is similar to the LMA-ProSealTM, whether the position of the air-QⓇ in relation to the vocal cords, as assessed by fiberoptic endoscopy, is similar to that of the LMA-ProSealTM and whether airway morbidity is similar between the air-QⓇ and the LMA-ProSealTM.

DETAILED DESCRIPTION:
Introduction:

The air-QⓇ Intubating Laryngeal Airway (ILA) (Mercury Medical, Clearwater, Fl.) is a newer supraglottic airway. It is approved for use as a primary airway and as an aid for intubation in situations of anticipated or unanticipated difficult airways. A unique feature of this device as compared to other airways on the market is the size of the inner diameter (ID) and length of its airway tube. Direct placement of tracheal tubes > 7.5 mm ID through the airway tube is possible.

The ProSealTM LMA (LMA North America, La Jolla, CA) is considered the gold standard for supraglottic devices with respect to airway seal pressure. On average, it is reported to be approximately 28 cmH2O. This is significantly higher than that of the first generation LMA, the LMA-ClassicTM, which has a maximum seal pressure of 20 cmH2O, but averages 16-18 cmH2O in actual practice.

Pilot data from 50 insertions of the air-QⓇ at our institution places the device intermediate to the two aforementioned LMAs with regard to seal pressure, with a mean seal pressure of 23 (12-30) cmH2O.

Specific Aims:

1. To test whether the air-QⓇ creates an airway seal pressure that is similar to the LMA-ProSealTM.
2. To test whether the position of the air-QⓇ in relation to the vocal cords, as assessed by fiberoptic endoscopy, is similar to that of the LMA-ProSealTM.
3. To test whether airway morbidity is similar between the air-QⓇ and the LMA-ProSealTM

Study design:

Prospective, single-center, randomized, controlled trial

Methods:

The patient will be met in the pre-operative area by the attending anesthesiologist, who interviews and examines the patient. A full explanation of the general anesthetic, including risks and benefits, will be given and informed consent obtained. An intravenous catheter will be placed and patients will be premedicated as needed at the discretion of the attending anesthesiologist. In the operating room, the patient will undergo standard monitoring per established American Society of Anesthesiology (ASA) guidelines. After a period of breathing 100% oxygen by facemask, anesthesia will be induced intravenously typically with fentanyl 0.5-1.5 mcg.kg -1 (a fast acting narcotic) and propofol (a potent sedative/amnestic agent) 2-3 mg.kg -1. After eyelash reflex is lost (i.e. the patient is asleep and not breathing), the patient will typically be ventilated with a facemask to demonstrate the patency of the airway. The LMA will then be placed using a standard technique. The cuff of the LMA will be inflated and the adequacy of placement assessed by presence of end-tidal carbon dioxide and adequate chest rise. The airway seal pressure will then be assessed by closing the APL valve on the anesthesia machine with a fresh gas flow of 5 liters/minute until an audible leak is observed. A stethoscope will be placed over the stomach while the valve is closed to listen for gastric insufflation. Administration of other anesthetic medication or muscle relaxants is at the discretion of the anesthesiologist and based on their clinical judgment and/or at the request of the surgeon. The anesthesia provider will not be blinded and will have access to all the monitors. The study deviates from routine care in that the choice of which LMA to use will be randomized by opening a sealed envelope prior to the start of the case. In addition, once the LMA has been placed and secured and the patient is stable from an anesthetic point of view, a flexible fiberoptic camera will be place into the airway tube of the LMA and the view of the patient's vocal cords in relation to the cuff of the LMA will be assessed.

At the conclusion of the case, when the patient is breathing on their own and is awake enough, as judged by the anesthesia provider, the LMA will be removed, as would be otherwise done as standard of care. The study LMA will be examined by a data collector for the presence of grossly visible blood or bile, and its presence or absence will be recorded. In the recovery area, once the patient is fully awake, as judged by the recovery staff, an observer will administer a standard oral questionnaire to the patient to determine if a sore throat, difficulty swallowing, or difficulty speaking is present. The patient will be called 24 hours later by the data collector and the same questionnaire will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or greater may be included if they presenting for any elective surgery or procedure to take place in any anesthetic location and require placement of a LMA for their surgery or procedure.

Exclusion Criteria:

* non-English speaking
* pregnant
* are a minor
* are a prisoner
* have impaired decision-making capacity or any condition for which the primary anesthesia team deems intubation with a tracheal tube to be necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher M Schroeder, MD, Principal Investigator — University of Wisconsin School of Medicine and Public Health Department of Anesthesiology
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Background] Cook TM, Lee G, Nolan JP. The ProSeal laryngeal mask airway: a review of the literature. Can J Anaesth. 2005 Aug-Sep;52(7):739-60. doi: 10.1007/BF03016565. PMID 16103390
- [Background] Wong DT, McGuire GP. Endotracheal intubation through a laryngeal mask/supraglottic airway. Can J Anaesth. 2007 Jun;54(6):489-91; author reply 491. doi: 10.1007/BF03022042. No abstract available. PMID 17541083

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Air-Q LMA | Proseal LMA
Started | 52 | 48
Completed | 52 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air-Q LMA | Proseal LMA | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 51 | 45 | 96
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (12) | 39 (14) | 39 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 28 | 25 | 53
Region of Enrollment [Number; unit: participants]
  United States | 52 | 48 | 100

OUTCOME MEASURES:

1. Primary Outcome: Airway Seal Pressure
Description: The airway seal pressure will then be assessed by closing the APL valve on the anesthesia machine with a fresh gas flow of 5 liters/minute until an audible leak is observed.
Time Frame: Intraoperative (day 1)
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Air-Q LMA | Proseal LMA
Number analyzed (Participants) | 52 | 48
cmH2O | 30 (7) | 30 (6)

2. Secondary Outcome: Grossly Visible Blood or Bile on LMA
Description: At the conclusion of the case, when the patient is breathing on their own and is awake enough, as judged by the anesthesia provider, the LMA will be removed, as would be otherwise done as standard of care. The study LMA will be examined by a data collector for the presence of grossly visible blood or bile, and its presence or absence will be recorded.
Time Frame: Upon LMA removal
Measure: Number; unit: participants
Arm/Group | Air-Q LMA | Proseal LMA
Number analyzed (Participants) | 52 | 48
participants | 10 | 4

3. Secondary Outcome: Glottic View
Description: Once the LMA has been placed and secured and the patient is stable from an anesthetic point of view, a flexible fiberoptic camera will be place into the airway tube of the LMA and the view of the patient's vocal cords in relation to the cuff of the LMA will be assessed.
Time Frame: Intraoperative (day 1)
Measure: Number; unit: participants with grade 1 glottic view
Arm/Group | Air-Q LMA | Proseal LMA
Number analyzed (Participants) | 52 | 48
participants with grade 1 glottic view | 41 | 29

4. Secondary Outcome: Airway Pathology
Description: In the recovery area, once the patient is fully awake, as judged by the recovery staff, an observer will administer a standard oral questionnaire to the patient to determine if a sore throat is present.
Time Frame: Postoperative (day 1) in recovery room
Measure: Number; unit: participants
Arm/Group | Air-Q LMA | Proseal LMA
Number analyzed (Participants) | 52 | 48
participants | 24 | 18

5. Secondary Outcome: Airway Pathology
Description: The patient will be called 24 hours later by the data collector who will administer a standard oral questionnaire to the patient to determine if a sore throat is present.
Time Frame: Postoperative Day Two
Measure: Number; unit: participants
Arm/Group | Air-Q LMA | Proseal LMA
Number analyzed (Participants) | 43 | 39
participants | 21 | 10

ADVERSE EVENTS:
Arm/Group | Air-Q LMA | Proseal LMA
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/48
Other Adverse Events (participants affected / at risk) | 0/52 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes